CLINICAL TRIAL: NCT05578976
Title: A Phase 3, Randomized, Open-Label Study to Evaluate Safety and Efficacy of Epcoritamab in Combination With R-CHOP Compared to R-CHOP in Subjects With Newly Diagnosed Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: A Study to Evaluate Change in Disease Activity of Subcutaneous (SC) Epcoritamab Combined With Intravenous and Oral Rituximab, Cyclophosphamide, Doxorubicin Hydrochloride, Vincristine, and Prednisone (R-CHOP) or R-CHOP in Adult Participants With Newly Diagnosed Diffuse Large B-Cell Lymphoma (DLBCL)
Acronym: EPCORE DLBCL-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M20-621; 2023-505277-32 (Other: EU CT)
Record Dates: First submitted 2022-10-12; First posted 2022-10-13 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: Relapsed or Refractory Diffuse Large B-Cell Lymphoma; Non-Hodgkins Lymphoma; Cancer; Epcoritamab; ABBV-GMAB-3013; R-CHOP; Rituximab; EPCORE
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence; Lymphoma, Non-Hodgkin; Neoplasms | interventions — Cyclophosphamide; Rituximab; Vincristine; Doxorubicin; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Epcoritamab and R-CHOP (Experimental): Participants will receive subcutaneous epcoritamab combined with intravenous rituximab, cyclophosphamide, doxorubixin hydrochloride, vincristine and oral prednisone (R-CHOP) followed by epcoritamab in 21-day cycles.
  Interventions: Drug: Epcoritamab; Drug: Cyclophosphamide; Drug: Rituximab; Drug: Vincristine; Drug: Doxorubicin; Drug: Prednisone
- R-CHOP and Rituximab (Experimental): Participants will receive intravenous rituximab, cyclophosphamide, doxorubixin hydrochloride, vincristine and oral prednisone (R-CHOP) followed by intravenous rituximab in 21-day cycles.
  Interventions: Drug: Cyclophosphamide; Drug: Rituximab; Drug: Vincristine; Drug: Doxorubicin; Drug: Prednisone

INTERVENTIONS:
Drug: Epcoritamab — Subcutaneous Injection (SC)
  Other Names: ABBV-GMAB-3013
  Arms: Epcoritamab and R-CHOP
Drug: Cyclophosphamide — Intravenous (IV) Injection
Drug: Rituximab — IV Infusion
Drug: Vincristine — IV Infusion
Drug: Doxorubicin — IV Infusion
Drug: Prednisone — Oral; Tablet

SUMMARY:
B-cell Lymphoma is an aggressive and rare cancer of a type of immune cells (a white blood cell responsible for fighting infections). The purpose of this study is to assess the change in disease activity of epcoritamab when combined with intravenous and oral rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine, and prednisone (R-CHOP) or R-CHOP in adult participants globally with diffuse large b-cell lymphoma (DLBCL). Change in disease activity will be assessed.

Epcoritamab is an investigational drug being developed for the treatment of DLBCL. Study doctors put the participants in groups called treatment arms. Participants will receive epcoritamab combined with R-CHOP, followed by epcoritamab or R-CHOP followed by rituximab will be explored. Approximately 900 adult participants with with newly diagnosed DLBCL will be enrolled in the study in approximately 315 sites in globally.

In the Arm 1, participants will receive subcutaneous epcoritamab combined with intravenous and oral R-CHOP followed by subcutaneous epcoritamab in 21-day cycles. In the Arm 2, participants will receive intravenous and oral R-CHOP followed by intravenous rituximab in 21-day cycles.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at an approved institution (hospital or clinic). The effect of the treatment will be frequently checked by medical assessments, blood tests, questionnaires and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Planned to receive treatment with 6 cycles of standard rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine, and prednisone (R-CHOP) per investigator determination.
* Must have newly diagnosed, histologically confirmed CD20+ diffuse large b-cell lymphoma [DLBCL] (de novo or histologically transformed from a diagnosis of follicular lymphoma) at most recent representative tumor biopsy based on the pathology report, with a World Health Organization (WHO) 2016 classification and including:

  * DLBCL, Not Otherwise Specified (NOS).
  * High grade B-cell lymphoma with MYC and BCL-2 and/or BCL-6 rearrangement with DLBCL morphology.
  * T-cell/histiocyte-rich large B-cell lymphoma.
  * Epstein Barr virus-positive DLBCL, NOS.
  * Follicular lymphoma Grade 3b.

Note: The local pathology report must be available at Screening to support CD20+ DLBCL histology.

Composite/intermediate histology with any of the following components is not allowed: high grade B-cell lymphoma, NOS; Hodgkin's lymphoma; primary mediastinal (thymic) large B-cell lymphoma; Burkitt; plasmablastic lymphoma or any CD20- lymphoma, such as anaplastic lymphoma kinase-positive large B-cell lymphoma, human herpesvirus type 8-positive DLBCL, or primary effusion lymphoma.

* Availability of archival or fresh or paraffin embedded tissue at Screening.
* Must have an IPI score of 2-5. The number of participants with IPI 2 will not exceed approximately 30% of the overall sample size.
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2 prior to initiating R-CHOP treatment. Note that participant with an initial ECOG performance status >= 3 may be screened if pre-phase treatment is planned. Participant may be eligible if ECOG performance status were to improve to 0-2 during pre-phase treatment.
* Has at least one target lesion defined as:

  * >= 1 measurable nodal lesion (long axis > 1.5 cm ) or >= 1 measurable extra-nodal lesion (long axis > 1 cm) on computed tomography (CT) scan or magnetic resonance imaging (MRI). AND
  * Positron emission tomography (PET)-positive on PET-CT scan.
* Laboratory values meeting the criteria laid out in the protocol.
* Left ventricular ejection fraction must be >= 50% by multi-gated acquisition or transthoracic echocardiography at Screening.

Exclusion Criteria:

* History of prior systemic anti-lymphoma therapy for diagnosed diffuse large b-cell lymphoma (DLBCL) including any definitive radiotherapy with curative intent] other than corticosteroids with or without vincristine during prephase treatment, or non-curative intent palliative radiotherapy with the stipulation that radiated lesions cannot be selected as target lesion for response assessment.
* Clinically significant cardiovascular disease as per the protocol.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Progression-Free Survival (PFS) with an International Prognostic Index (IPI) of 3-5 | Up to Approximately 46 Months
  PFS is defined as the duration from randomization to the date of disease progression as determined by Lugano 2014 criteria as assessed by Independent Review Committee (IRC), or death due to any cause whichever comes first.

SECONDARY OUTCOMES:
Number of Participants with PFS | Up to Approximately 46 Months
  PFS is defined as the duration from randomization to the date of disease progression as determined by Lugano 2014 criteria as assessed by IRC, or death due to any cause, whichever occurs first.
Number of Participants with Event-free survival (EFS) | Up to Approximately 46 Months
  EFS is defined as the duration from randomization to the date of disease progression determined by Lugano criteria as assessed by IRC, IRC-assessed PR or SD followed by non protocol-specified NALT, a positive biopsy on or after end-of-treatment (EOT), regardless of whether NAL initiated, or death from any cause.
Percentage of Participants with Complete Remission (CR) | On or After to Approximately 28 Weeks
  CR on or after EOT, determined by Lugano 2014 criteria as assessed by IRC.
Overall survival (OS) | Up to Approximately 76 Months
  OS is defined as time from randomization until death due to any causes.
Percentage of Participants with Minimal Residual Disease (MRD) Negativity | Up to Approximately 46 Months
  The MRD negativity rate is defined as the percentage of participants who achieve MRD negativity prior to the initiation of any non-protocol-specified new anti-lymphoma therapy.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (331):
- United States (68):
  - University of Arizona Cancer Center - North Campus /ID# 227463, Tucson, Arizona
  - Yuma Regional Medical Center /ID# 261527, Yuma, Arizona
  - University of Arkansas for Medical Sciences /ID# 225703, Little Rock, Arkansas
  - CBCC Global Research, Inc. /ID# 262037, Bakersfield, California
  - Alta Bates Summit Medical Center for Research /ID# 229427, Berkeley, California
  - Orange Coast Memorial Medical Center /ID# 229632, Fountain Valley, California
  - Providence - St. Jude Medical Center /ID# 262042, Fullerton, California
  - Saddleback Memorial Medical Center /ID# 229631, Laguna Hills, California
  - Long Beach Memorial Medical Ct /ID# 228996, Long Beach, California
  - Cancer and Blood Speciality Clinic - Los Alamitos /ID# 262032, Los Alamitos, California
  - University of Southern California /ID# 225443, Los Angeles, California
  - University of California, Los Angeles /ID# 226887, Los Angeles, California
  - Kaiser Permanente, Waterpark III Institute for Health Research /ID# 228618, Aurora, Colorado
  - Cancer Specialists of North Florida /ID# 226826, Jacksonville, Florida
  - Ocala Oncology Florida Cancer Affiliates - Main /ID# 262785, Ocala, Florida
  - Orlando Health Cancer Institute /ID# 232626, Orlando, Florida
  - Straub Medical Center /ID# 229464, Honolulu, Hawaii
  - University of Illinois at Chicago /ID# 226889, Chicago, Illinois
  - Southern IL Univ School of Med /ID# 228999, Springfield, Illinois
  - Springfield Clinic Main Campus /ID# 262584, Springfield, Illinois
  - Carle Cancer Institute /ID# 228338, Urbana, Illinois
  - Parkview Comprehensive Cancer Center /ID# 227026, Fort Wayne, Indiana
  - Goshen Center for Cancer Care /ID# 225534, Goshen, Indiana
  - University of Iowa Health Care /ID# 261945, Des Moines, Iowa
  - Cancer Center of Kansas /ID# 261983, Wichita, Kansas
  - Norton Cancer Institute - St. Matthews /ID# 225420, Louisville, Kentucky
  - University of Maryland, Baltimore /ID# 225421, Baltimore, Maryland
  - Johns Hopkins Hospital /ID# 225369, Baltimore, Maryland
  - American Oncology Partners of Maryland /ID# 226859, Bethesda, Maryland
  - UMass Memorial Medical Center /ID# 226939, Worcester, Massachusetts
  - University of Michigan Comprehensive Cancer Center Michigan Medicine /ID# 225462, Ann Arbor, Michigan
  - Trinity Health St. Joseph Mercy Ann Arbor /ID# 228206, Ypsilanti, Michigan
  - Metro Minnesota Community Oncology Research Consortium (MMCORC) /ID# 226680, Saint Louis Park, Minnesota
  - University of Mississippi Medical Center /ID# 228045, Jackson, Mississippi
  - Intermountain Health St. Vincent Regional Hospital - Cancer Centers of Montana /ID# 259014, Billings, Montana
  - NHO Revive Research Institute, LLC /ID# 261113, Lincoln, Nebraska
  - MDACC Cooper /ID# 260320, Camden, New Jersey
  - Titan Health Partners LLC, d/b/a Astera Cancer Care /ID# 226654, East Brunswick, New Jersey
  - Morristown Medical Center /ID# 239457, Morristown, New Jersey
  - University of New Mexico /ID# 227332, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital /ID# 262084, Albuquerque, New Mexico
  - Presbyterian Rust Medical Center /ID# 262068, Rio Rancho, New Mexico
  - Roswell Park Cancer Institute /ID# 239127, Buffalo, New York
  - NYU Langone Hospital - Long Island /ID# 262412, Mineola, New York
  - New York Cancer and Blood Specialists- New Hyde Park /ID# 265392, New Hyde Park, New York
  - NYU Langone - Laura and Isaac Perlmutter Cancer Center /ID# 226141, New York, New York
  - New York Cancer and Blood Specialists- Manhattan /ID# 265391, New York, New York
  - Icahn School of Medicine at Mount Sinai /ID# 225370, New York, New York
  - Memorial Sloan Kettering Cancer Center-Koch Center /ID# 225379, New York, New York
  - New York Cancer and Blood Specialists /ID# 261114, Port Jefferson Station, New York
  - New York Cancer and Blood Specialists- Eastchester, Bronx /ID# 265396, The Bronx, New York
  - Novant Health Presbyterian Medical Center /ID# 227753, Charlotte, North Carolina
  - East Carolina University - Brody School of Medicine /ID# 225992, Greenville, North Carolina
  - Novant Health Forsyth Medical Center /ID# 228339, Winston-Salem, North Carolina
  - University of Cincinnati /ID# 225374, Cincinnati, Ohio
  - OhioHealth Arthur G.H. Bing, MD Cancer Center /ID# 260790, Columbus, Ohio
  - University of Oklahoma, Stephenson Cancer Center /ID# 225556, Oklahoma City, Oklahoma
  - Kaiser Permanente - Northwest /ID# 225488, Portland, Oregon
  - Houston Methodist Hospital /ID# 258957, Houston, Texas
  - Millennium Research & Clinical Development /ID# 228284, Kingwood, Texas
  - Joe Arrington Cancer Research /ID# 227217, Lubbock, Texas
  - Baylor Scott & White Medical Center- Temple /ID# 225935, Temple, Texas
  - Intermountain Medical Center /ID# 231184, Murray, Utah
  - University of Virginia Cancer Center - West Complex /ID# 225433, Charlottesville, Virginia
  - Virginia Commonwealth University Medical Center Main Hospital /ID# 225796, Richmond, Virginia
  - Vista Oncology - East Olympia /ID# 229375, Olympia, Washington
  - MultiCare Institute for Research & Innovation /ID# 225432, Tacoma, Washington
  - MultiCare Regional Cancer Center - Tacoma /ID# 265285, Tacoma, Washington
- Australia (8):
  - Liverpool Hospital /ID# 230072, Liverpool, New South Wales
  - Royal Adelaide Hospital /ID# 225683, Adelaide, South Australia
  - Monash Health - Monash Medical Centre /ID# 225680, Clayton, Victoria
  - Austin Health /ID# 225716, Heidelberg, Victoria
  - The Alfred Hospital /ID# 225999, Melbourne, Victoria
  - Hollywood Private Hospital /ID# 251837, Nedlands, Western Australia
  - Perth Blood Institute Ltd /ID# 225679, Nedlands, Western Australia
  - Royal Perth Hospital /ID# 226583, Perth, Western Australia
- Austria (4):
  - Universitaetsklinikum St. Poelten /ID# 234016, Sankt Pölten, Lower Austria
  - Medizinische Universitaet Wien /ID# 252095, Vienna, Vienna
  - Klinik Ottakring /ID# 243941, Vienna, Vienna
  - Landeskrankenhaus Salzburg-Universitaetsklinikum der PMU (LKH) /ID# 228360, Salzburg
- Belgium (12):
  - Duplicate_ZAS Middelheim /ID# 225741, Antwerp, Antwerpen
  - ZAS Cadix /ID# 264327, Antwerp, Antwerpen
  - Cliniques Universitaires UCL Saint-Luc /ID# 225737, Woluwe-Saint-Lambert, Brussels Capital
  - Hospital La Louviere Site Jolimont - Helora /ID# 225738, La Louvière, Hainaut
  - CHU de Liège /ID# 225952, Liège, Liege
  - Université Catholique de Louvain-Namur - Centre Hospitalier Universitaire Dinant /ID# 225742, Yvoir, Namur
  - UZ Gent /ID# 250031, Ghent, Oost-Vlaanderen
  - Vitaz /Id# 226153, Sint-Niklaas, Oost-Vlaanderen
  - Universitair Ziekenhuis Leuven /ID# 225951, Leuven, Vlaams-Brabant
  - AZ-Delta /ID# 225736, Roeselare, West-Vlaanderen
  - Institut Jules Bordet /ID# 225954, Anderlecht
  - AZ Sint-Jan Brugge /ID# 225735, Bruges
- Brazil (10):
  - Hospital de Clinicas da Universidade Federal do Parana /ID# 226027, Curitiba, Paraná
  - Hospital Erasto Gaertner /ID# 262593, Curitiba, Puerto Rico
  - Hospital Amaral Carvalho - Fundacao Doutor Amaral Carvalho /ID# 226065, Jaú, São Paulo
  - Fundacao Antonio Prudente - AC Camargo Cancer Center /ID# 226809, São Paulo, São Paulo
  - Sociedade Beneficente Israelita Brasileira Hospital Albert Einstein /ID# 252832, São Paulo, São Paulo
  - Instituto Nacional de Cancer (INCA) /ID# 226026, Rio de Janeiro
  - Real e Benemérita Associação Portuguesa de Beneficência /ID# 226023, São Paulo
  - Hospital Alemao Oswaldo Cruz /ID# 252833, São Paulo
  - Instituto D'Or de Pesquisa e Ensino - Regional Sao Paulo /ID# 262394, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao /ID# 226048, São Paulo
- Bulgaria (4):
  - UMHAT Sveti Georgi /ID# 245780, Plovdiv
  - Acibadem City Clinic Tokuda University Hospital EAD /ID# 244616, Sofia
  - UMHAT Sveti Ivan Rilski /ID# 244615, Sofia
  - SHAT Hematologic Diseases /ID# 250102, Sofia
- Canada (5):
  - Arthur J.E. Child Comprehensive Cancer Centre Pharmacy /ID# 226077, Calgary, Alberta
  - BC Cancer - Vancouver /ID# 230573, Vancouver, British Columbia
  - William Osler Health System /ID# 250973, Brampton, Ontario
  - Juravinski Cancer Centre /ID# 226084, Hamilton, Ontario
  - Saskatoon Cancer Centre /ID# 226082, Saskatoon, Saskatchewan
- China (27):
  - The Fifth Medical Center of PLA General Hospital /ID# 230941, Beijing, Beijing Municipality
  - Beijing Cancer Hospital /ID# 229819, Beijing, Beijing Municipality
  - Peking University Third Hospital /ID# 230975, Beijing, Beijing Municipality
  - Fujian Provincial Cancer Hospital /ID# 238430, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University /ID# 238426, Xiamen, Fujian
  - Sun Yat-Sen University Cancer Center /ID# 238371, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital /ID# 230945, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University /ID# 238436, Guangzhou, Guangdong
  - Fourth Hospital of Hebei Medical University /ID# 238656, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital /Id# 241755, Harbin, Heilongjiang
  - Henan Cancer Hospital /ID# 230398, Zhengzhou, Henan
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Sc /ID# 234152, Wuhan, Hubei
  - Hubei Cancer Hospital /ID# 232256, Wuhan, Hubei
  - The First Affiliated Hospital of Soochow University /ID# 232569, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical College /ID# 233174, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University /ID# 230399, Nanchang, Jiangxi
  - Jiangxi Provincial Cancer Hospital /ID# 233379, Nanchang, Jiangxi
  - The First Hospital of Jilin University /ID# 239618, Changchun, Jilin
  - The First Hospital of China Medical University /ID# 233201, Shenyang, Liaoning
  - Shandong Cancer Hospital /ID# 233200, Jinan, Shandong
  - Fudan University Cancer Hospital /ID# 251516, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital /ID# 250745, Taiyuan, Shanxi
  - Tianjin Cancer Hospital /ID# 230974, Tianjin, Tianjin Municipality
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sc /ID# 259904, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine /ID# 230387, Hangzhou, Zhejiang
  - The second affiliated hospital of Zhejiang University school of medicine /ID# 231249, Hangzhou, Zhejiang
  - Zhejiang Cancer hospital /ID# 231388, Hangzhou, Zhejiang
- Croatia (6):
  - Clinical Hospital Dubrava /ID# 251809, Zagreb, City of Zagreb
  - Klinicka bolnica Merkur /ID# 252481, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Zagreb /ID# 250709, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Rijeka /ID# 251811, Rijeka, Primorje-Gorski Kotar County
  - Klinicki Bolnicki Centar (KBC) Split /ID# 250729, Split, Split-Dalmatia County
  - Opca bolnica Dr. Josip Bencevic /ID# 251812, Slavonski Brod
- Czechia (6):
  - Fakultní Nemocnice Brno - Jihlavská /ID# 225953, Brno, Brno-mesto
  - Fakultní nemocnice Hradec Králové - Sokolská /ID# 225955, Hradec Králové, Hradec Kralove
  - Fakultni Nemocnice Ostrava /ID# 225957, Ostrava, Ostrava-mesto
  - Fakultni nemocnice Kralovske Vinohrady /ID# 225956, Prague
  - Vseobecna fakultni nemocnice v Praze /ID# 225396, Prague
  - Duplicate_Fakultni Nemocnice v Motole /ID# 225958, Prague
- Denmark (5):
  - Rigshospitalet /ID# 226576, Copenhagen Ø, Capital Region
  - Aarhus Universitetshospital - Skejby /ID# 226594, Aarhus, Central Jutland
  - Roskilde Sygehus /ID# 226597, Roskilde, Region Sjælland
  - Odense University Hospital /ID# 226593, Odense, Region Syddanmark
  - Sygehus Lillebalt, Vejle /ID# 226592, Vejle, Region Syddanmark
- France (23):
  - CHU de Nice - Hôpital Archet 1 /ID# 226127, Nice, Alpes-Maritimes
  - CHU Clermont-Ferrand /ID# 229283, Clermont, Auvergne-Rhône-Alpes
  - Institut Paoli-Calmettes /ID# 226557, Marseille, Bouches-du-Rhone
  - CHU de Rennes - PONTCHAILLOU /ID# 228207, Rennes, Brittany Region
  - CHU Dijon /ID# 238345, Dijon, Cote-d Or
  - CHU Limoges - Dupuytren 1 /ID# 234235, Limoges, Franche-Comte
  - CHU Montpellier - Hopital Saint Eloi /ID# 228191, Montpellier, Herault
  - CHU Grenoble - Hopital Michallon /ID# 226128, La Tronche, Isere
  - CHRU Nancy - Hopitaux de Brabois /ID# 226102, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - CHRU Lille - Hopital Claude Huriez /ID# 226101, Lille, Nord
  - Hopitaux Universitaires Henri Mondor - Hopital Henri Mondor /ID# 226560, Créteil, Paris
  - CHU de Nantes, Hotel Dieu -HME /ID# 226125, Nantes, Pays de la Loire Region
  - Centre Hospitalier de la Cote Basque /ID# 249143, Bayonne, Pyrenees-Atlantiques
  - HCL - Hopital Lyon Sud /ID# 227086, Pierre-Bénite, Rhone
  - Centre Henri Becquerel /ID# 226103, Rouen, Seine-Maritime
  - CHU Amiens-Picardie Site Sud /ID# 238347, Amiens, Somme
  - CHD Vendée- La Roche-sur-Yon - Les Oudairies /ID# 243899, La Roche-sur-Yon, Vendee
  - CHU Poitiers - La miletrie /ID# 226578, Poitiers, Vienne
  - Chu Angers /Id# 245931, Angers
  - CHU de CAEN - Hopital de la Cote de Nacre /ID# 226582, Caen
  - Hôpital Saint-Louis /ID# 226126, Paris
  - Institut Curie - site CLCC René Huguenin /ID# 253519, Saint-Cloud
  - Hopital Pitie Salpetriere /ID# 238343, Paris, Île-de-France Region
- Greece (7):
  - General Hospital of Athens Laiko /ID# 225399, Athens, Attica
  - Alexandra General Hospital /ID# 225402, Athens, Attica
  - University General Hospital Attikon /ID# 225401, Athens, Attica
  - General Hospital of Athens Evaggelismos and Ophthalmiatrio of Athens Polyclinic /ID# 225416, Athens
  - University General Hospital of Ioannina /ID# 225400, Ioannina
  - General University Hospital of Thessaloniki AXEPA /ID# 225398, Thessaloniki
  - Theageneio Anticancer Hospital /ID# 225516, Thessaloniki
- Hungary (8):
  - Gyor-Moson-Sopron Varmegyei Petz Aladar Egyetemi Oktato Korhaz /ID# 257189, Győr, Győr-Moson-Sopron
  - Debreceni Egyetem-Klinikai Kozpont /ID# 226821, Debrecen, Hajdú-Bihar
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz /ID# 245938, Kaposvár, Somogy County
  - Tolna Varmegyei Balassa Janos Korhaz /ID# 250063, Szekszárd, Tolna County
  - Vas Varmegyei Markusovszky Egyetemi Oktatokorhaz /ID# 226846, Szombathely, Vas County
  - Semmelweis Egyetem /ID# 227239, Budapest
  - Orszagos Onkologiai Intezet /ID# 227294, Budapest
  - Szegedi Tudományegyetem /ID# 226838, Szeged
- Israel (8):
  - Meir Medical Center /ID# 225612, Kfar Saba, Central District
  - Assuta Tel Aviv Medical Center /ID# 226066, Tel Aviv, Central District
  - Rambam Health Care Campus /ID# 225981, Haifa, H_efa
  - Shaare Zedek Medical Center /ID# 259796, Jerusalem, Jerusalem
  - Hadassah /ID# 225614, Jerusalem, Jerusalem
  - The Chaim Sheba Medical Center /ID# 225600, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 225891, Tel Aviv, Tel Aviv
  - Rabin Medical Center /ID# 225862, Petah Tikva
- Italy (16):
  - IRCCS AOU di Bologna - Policlinico Sant'Orsola-Malpighi /ID# 225551, Bologna, Emilia-Romagna
  - Fondazione di Religione e di Culto Casa Sollievo della Sofferenza /ID# 225554, San Giovanni Rotondo, Foggia
  - IRCCS Ospedale San Raffaele /ID# 225555, Milan, Milano
  - Istituto Europeo Di Oncologia /ID# 225545, Milan, Milano
  - Azienda Ospedaliera Universitaria Federico II /ID# 225543, Naples, Napoli
  - A.O.U. CITTA' DELLA SALUTE E DELLA SCIENZA DI TORINO - Ospedale Molinette /ID# 225775, Turin, Piedmont
  - Duplicate_Centro di Riferimento Oncologico /ID# 225553, Aviano, Pordenone
  - Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST - IRCCS /ID# 252192, Meldola, Reggio Emilia
  - Istituto di Candiolo Fondazione del Piemonte per l'Oncologia IRCCS /ID# 225751, Candiolo, Torino
  - Azienda Ospedaliero - Universitaria SS. Antonio e Biagio e Cesare Arrigo - Aless /ID# 225542, Alessandria
  - I.R.C.C.S Istituto Tumori Giovanni Paolo II /ID# 225548, Bari
  - Duplicate_ASST Spedali civili di Brescia /ID# 225549, Brescia
  - Azienda Ospedaliero Universitaria Maggiore della Carita di Novara /ID# 225773, Novara
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello /ID# 225541, Palermo
  - Azienda Ospedaliero Universitaria Pisana /ID# 225575, Pisa
  - Ospedale Santa Maria Delle Croci /ID# 225571, Ravenna
- Japan (20):
  - NHO Nagoya Medical Center /ID# 230677, Nagoya, Aichi-ken
  - Aichi Cancer Center Hospital /ID# 226090, Nagoya, Aichi-ken
  - National Cancer Center Hospital East /ID# 250151, Kashiwa-shi, Chiba
  - Matsuyama Red Cross Hospital /ID# 251068, Matsuyama, Ehime
  - National Hospital Organization Kyushu Cancer Center /ID# 251622, Fukuoka, Fukuoka
  - Kyushu University Hospital /ID# 226091, Fukuoka, Fukuoka
  - Fukushima Medical University Hospital /ID# 250869, Fukushima, Fukushima
  - Duplicate_Hokkaido University Hospital /ID# 250149, Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital /ID# 250597, Kobe, Hyōgo
  - University of Tsukuba Hospital /ID# 251282, Tsukuba, Ibaraki
  - Kanazawa University Hospital /ID# 251770, Kanazawa, Ishikawa-ken
  - Kagoshima University Hospital /ID# 250163, Kagoshima, Kagoshima-ken
  - Tokai University Hospital /ID# 251281, Isehara, Kanagawa
  - Tohoku University Hospital /ID# 250150, Sendai, Miyagi
  - Okayama University Hospital /ID# 250161, Okayama, Okayama-ken
  - Kindai University Hospital /ID# 250160, Osakasayama-shi, Osaka
  - Osaka University Hospital /ID# 251283, Suita-shi, Osaka
  - National Cancer Center Hospital /ID# 226089, Chuo-ku, Tokyo
  - The Cancer Institute Hospital Of JFCR /ID# 230269, Koto-ku, Tokyo
  - Yamagata University Hospital /ID# 230003, Yamagata, Yamagata
- Netherlands (26):
  - Flevo Ziekenhuis /ID# 229606, Almere Stad, Flevoland
  - Gelre Ziekenhuizen /ID# 229762, Apeldoorn, Gelderland
  - Canisius-Wilhelmina Ziekenhuis /ID# 231291, Nijmegen, Gelderland
  - Maastricht Universitair Medisch Centrum /ID# 225607, Maastricht, Limburg
  - Amphia Ziekenhuis /ID# 229550, Breda, North Brabant
  - Catharina Ziekenhuis /ID# 230465, Eindhoven, North Brabant
  - Maxima Medisch Centrum /ID# 225603, Eindhoven, North Brabant
  - Elisabeth Tweesteden Ziekenhuis /ID# 229773, Tilburg, North Brabant
  - Noordwest Ziekenhuisgroep /ID# 230613, Alkmaar, North Holland
  - Vrije Universiteit Medisch Centrum /ID# 225608, Amsterdam, North Holland
  - Olvg /Id# 229761, Amsterdam, North Holland
  - Spaarne Gasthuis, Haarlem Zuid /ID# 229621, Haarlem, North Holland
  - Tergooi /ID# 229772, Hilversum, North Holland
  - Dijklander Ziekenhuis /ID# 229900, Hoorn, North Holland
  - Zaans Medisch Centrum /ID# 230614, Zaandam, North Holland
  - Medisch Spectrum Twente /ID# 225610, Enschede, Overijssel
  - Medisch Centrum Leeuwarden /ID# 225605, Leeuwarden, Provincie Friesland
  - Albert Schweitzer Ziekenhuis /ID# 229560, Dordrecht, South Holland
  - Leids Universitair Medisch Centrum /ID# 225606, Leiden, South Holland
  - Meander Medisch Centrum /ID# 229608, Amersfoort, Utrecht
  - St. Antonius Ziekenhuis /ID# 229901, Nieuwegein, Utrecht
  - Jeroen Bosch Ziekenhuis /ID# 229765, 's-Hertogenbosch
  - Deventer Ziekenhuis /ID# 229937, Deventer
  - Universitair Medisch Centrum Groningen /ID# 225602, Groningen
  - Haaglanden Medisch Centrum /ID# 229686, The Hague
  - Diakonessenhuis /ID# 251793, Utrecht
- New Zealand (2):
  - North Shore Hospital /ID# 250992, Takapuna, Auckland
  - Christchurch Hospital /ID# 250993, Christchurch, Canterbury
- Poland (5):
  - ARS-MEDICAL Sp. z o.o. /ID# 225848, Piła, Greater Poland Voivodeship
  - Centrum Medyczne Pratia Poznan /ID# 227236, Skórzewo, Greater Poland Voivodeship
  - Wojewodzki Szpital Specjalistyczny im. Janusza Korczaka /ID# 228723, Słupsk, Pomeranian Voivodeship
  - Szpital Kliniczny MSWiA z Warminsko-Mazurskim Centrum Onkologii /ID# 225985, Olsztyn, Warmian-Masurian Voivodeship
  - Swietokrzyskie Centrum Onkologii Samodzielny Publiczny Zaklad Opieki Zdrowotnej /ID# 225986, Kielce, Świętokrzyskie Voivodeship
- Portugal (4):
  - 2CA-Braga, Hospital de Braga /ID# 249112, Braga
  - IPO Lisboa FG, EPE /ID# 249109, Lisbon
  - Unidade Local de Saude de Santa Maria, EPE /ID# 249111, Lisbon
  - IPO Porto FG, EPE /ID# 249110, Porto
- Puerto Rico (2):
  - Hematology and Oncology Institute /ID# 230054, Manatí
  - Pan American Center for Oncology Trials, LLC /ID# 230052, Rio Piedras
- Slovakia (2):
  - Narodny onkologicky ustav /ID# 238847, Bratislava, Bratislava Region
  - Univerzitna nemocnica Martin /ID# 240828, Martin, Žilina Region
- South Africa (5):
  - Wits Clinical Research /ID# 227799, Johannesburg, Gauteng
  - Wits Clinical Research /ID# 227803, Johannesburg, Gauteng
  - Alberts Cellular Therapy /ID# 227798, Pretoria, Gauteng
  - University of Cape Town /ID# 227802, Cape Town, Western Cape
  - Haemalife Inc. /ID# 243391, Kuils River, Western Cape
- South Korea (10):
  - Inje University - Busan Paik Hospital /ID# 232262, Busan, Busan Gwang Yeogsi
  - Seoul National University Bundang Hospital /ID# 225763, Seongnam-si, Gyeonggido
  - Keimyung University Dongsan Hospital /ID# 232264, Daegu, Gyeongsangbuk-do
  - Dong-A University Medical Center /ID# 228451, Pusan, Gyeongsangnam-do
  - Jeonbuk National University Hospital /ID# 232263, Jeonju, Jeonrabugdo
  - Seoul National University Hospital /ID# 225760, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center /ID# 225758, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 225759, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St. Marys Hospital /ID# 225761, Seoul, Seoul Teugbyeolsi
  - Ulsan University Hospital /ID# 226971, Ulsan, Ulsan Gwang Yeogsi
- Spain (16):
  - Instituto Catalan de Oncologia (ICO) Badalona /ID# 228063, Badalona, Barcelona
  - Institut Català d'Oncologia (ICO) - L'Hospitalet /ID# 227393, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Reina Sofia /ID# 225806, Córdoba, Cordoba
  - Hospital Clinico Universitario Virgen de la Arrixaca /ID# 255381, El Palmar, Murcia
  - Clinica Universidad de Navarra - Pamplona /ID# 225809, Pamplona, Navarre
  - Hospital Parc de Salut del Mar /ID# 225810, Barcelona
  - Hospital Universitario Vall d'Hebron /ID# 225811, Barcelona
  - Hospital Clinic de Barcelona /ID# 226651, Barcelona
  - Hospital Santa Creu i Sant Pau /ID# 225813, Barcelona
  - CLINICA UNIVERSIDAD DE NAVARRA-Madrid /ID# 228228, Madrid
  - Hospital Universitario Infanta Leonor /ID# 225816, Madrid
  - MD Anderson Madrid /ID# 225817, Madrid
  - Hospital Universitario Ramon y Cajal /ID# 241750, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz /ID# 225804, Madrid
  - Hospital Universitario 12 de Octubre /ID# 225815, Madrid
  - Hospital Clinico Universitario de Valencia /ID# 225818, Valencia
- Sweden (5):
  - Skane University Hospital Lund /ID# 227285, Lund, Skåne County
  - Karolinska University Hospital Solna /ID# 229284, Solna, Stockholm County
  - Sodra Alvsborgs sjukhus /ID# 228885, Borås, Västra Götaland County
  - Sahlgrenska Universitetssjukhuset /ID# 250089, Gothenburg, Västra Götaland County
  - Linkoping University Hospital /ID# 233521, Linköping, Östergötland County
- Switzerland (3):
  - Kantonsspital Aarau AG /ID# 229112, Aarau, Canton of Aargau
  - Spital Thun /ID# 229499, Thun, Canton of Bern
  - KSW Kantonsspital Winterthur /ID# 241631, Winterthur, Canton of Zurich
- Taiwan (4):
  - Kaohsiung Chang Gung Memorial Hospital /ID# 226670, Kaohsiung City, Kaohsiung
  - China Medical University Hospital /ID# 226188, Taichung
  - Taichung Veterans General Hospital /ID# 226674, Taichung
  - National Cheng Kung University Hospital /ID# 226671, Tainan
- Turkey (Türkiye) (6):
  - Anadolu Saglik Merkezi /ID# 225777, Dilovası, Kocaeli
  - Ankara Universitesi Fakultesi /ID# 227331, Ankara
  - Inonu University Medical Faculty /ID# 226572, Malatya
  - Ondokuz Mayis Universitesi /ID# 251247, Samsun
  - Karadeniz University /ID# 226573, Trabzon
  - Baskent Universitesi Adana Uyg. ve Arast. Merkezi Yuregir Baskent Hastanesi /ID# 225921, Yüreğir
- United Kingdom (4):
  - Hammersmith Hospital /ID# 242215, London, England
  - Norfolk and Norwich University Hospitals NHS Foundation Trust /ID# 226692, Norwich, Norfolk
  - University Hospitals Birmingham NHS Foundation Trust /ID# 229197, Birmingham
  - NHS Lothian /ID# 229055, Edinburgh

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related info — https://www.abbvieclinicaltrials.com/study/?id=M23-362